CLINICAL TRIAL: NCT02629302
Title: Effects of Animal-assisted Therapy in Patients With Severe Disorders of Consciousness at REHAB Basel: a Randomised-controlled Trial
Brief Title: Effects of Animal Assisted Therapy on Patients With Severe Disorders of Consciousness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Institute for Interdisciplinary Research on the Human-Pet Relationship (Other); Rehab Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EKNZ 2015-153
Record Dates: First submitted 2015-12-07; First posted 2015-12-14 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2017-10

CONDITIONS: Disorder of Consciousness
MeSH Terms: conditions — Consciousness Disorders | interventions — Animal Assisted Therapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- animal assisted therapy (Experimental): "Standard" therapy (speech therapy, occupational therapy and physiotherapy) that is done in the presence and with Integration of an animal.
  Interventions: Other: animal assisted therapy
- standard therapy (Active Comparator): standard physiotherapy, standard speech therapy and standard occupational therapy
  Interventions: Other: standard therapy

INTERVENTIONS:
Other: animal assisted therapy — physiotherapy, speech therapy and occupational therapy in the presence of an animal
  Arms: animal assisted therapy
Other: standard therapy — standard physiotherapy, speech therapy and occupational therapy
  Arms: standard therapy

SUMMARY:
The study investigates the effects of animal-assisted therapy on patients with severe disorders of consciousness. The focus lies on the short-term biopsychosocial effects that occur when animals are present during therapy sessions in comparison to therapy sessions without animals, observing a group of 10 patients during 16 therapy sessions.

While half of the sessions are held in presence of an animal and half without, they are as comparable as possible with respect to content and setting. In this study, patients in a minimal conscious state are recruited.

DETAILED DESCRIPTION:
This pilot study is designed as a controlled cross-over, within-subject trial with repeated measurement. The experimental condition is the standardised therapy session using therapy animals (AAT), while the control condition is the comparable "standard" therapy session without the presence of an animal.

Over a period of four weeks, patients have four standardised therapy sessions per week, that alternate in a way that two sessions in two consecutive weeks are similar except for one is with the presence of animals and one without. In this way, data is collected over 16 therapy sessions (8 experimental, 8 control) for each patient.

Each therapy session lasts about 20 minutes.

The study takes place at REHAB Basel. Animal-assisted therapies are held in a special room at REHAB Basel in the presence of one or more small animals that will be selected by the therapist.

Patients are allocated randomly to start with either the experimental or the control condition.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients of REHAB Basel
* Disorder of consciousness: minimal conscious state defined via:
* CRS Score (Coma Remission Scale) of auditory 3-4 or visual 2-5 or motor 3-5 or oromotor/verbal = 3 or communication = 1
* BAVESTA Score of 2.8

Exclusion Criteria:

* Enrolment of the investigator, his/her family members, employees and other dependent persons
* medical contraindications for contact with animals as allergy, phobia etc.
* If the patient's medication changes radically during the time of data collection

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Degree of consciousness | 4 weeks
  assessed via behavioral coding in Noldus Observer

SECONDARY OUTCOMES:
Heart rate | 4 weeks
  assessed via non-invasive HR monitoring belts (Polar® RS800CX, Polar® Electro Oy)
Behavioral reaction | 4 weeks
  measured via therapist's ratings on the BAVESTA scale (Basler Assessment Vegetative State)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Hediger, Principal Investigator — Rehab Basel
Locations (1):
- REHAB Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hediger K, Petignat M, Marti R, Hund-Georgiadis M. Animal-assisted therapy for patients in a minimally conscious state: A randomized two treatment multi-period crossover trial. PLoS One. 2019 Oct 1;14(10):e0222846. doi: 10.1371/journal.pone.0222846. eCollection 2019. PMID 31574106